CLINICAL TRIAL: NCT02795338
Title: Multi-modality Localization of Eloquent Brain Function-A Comparison of Technologies for Improved Applicability
Brief Title: Multi-modality Localization of Eloquent Brain Function
Status: Withdrawn | Type: Observational
Why Stopped: Project did not receive funding and was never started
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0176-16-EP
Record Dates: First submitted 2016-05-24; First posted 2016-06-10 (Estimated); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms | interventions — Brain Mapping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: brain mapping — pre-operative and intra-operative brain mapping to identify eloquent areas

SUMMARY:
Accurate identification of areas of eloquent brain function is vital to surgical decision making and to preservation of independence as patients with brain tumors who are higher functioning have better survival outcomes. Eloquent brain is defined as a region controlling language, motor, or sensory function such that without its proper input, a person would be left with significant neurologic deficits. Imaging technology has evolved to provide multiple non-invasive modalities for pre-operative testing of eloquent brain function. Studies have shown that these non-invasive mapping modalities provide useful information, however, the information provided inconsistently predicts distribution of eloquent function.

Direct electrical stimulation (DES) at surgery allows assessment of eloquent function directly from the brain surface (invasive) and is considered the gold standard in brain mapping. Therefore, in order to determine the true clinical applicability of the non-invasive mapping technologies, this study proposes to assess the predictive value of functional MRI (fMRI) and magnetoencephalography (MEG) for sensorimotor and language functions by comparing results to DES and determine whether fMRI or MEG provides the most consistent and accurate information. The rationale for the proposed research is that understanding the reliability of our current technology will allow us to perform safer surgeries and to preserve neurologic function.

DETAILED DESCRIPTION:
It is unknown whether imaging technologies have broad applications in brain mapping due to limited knowledge of the value of the results. Accurate identification of areas of eloquent brain function is vital to surgical decision making and to preservation of independence as patients with brain tumors who are higher functioning have better survival outcomes. Imaging technology has evolved to provide multiple non-invasive modalities for pre-operative testing of eloquent brain function and include functional MRI (fMRI) and magnetoencephalography (MEG). Eloquent brain is defined as a region controlling language, motor, or sensory function such that without its proper input, a person would be left with significant neurologic deficits. Studies conducted have shown that these non-invasive mapping modalities provide useful information, however, the information provided inconsistently predicts distribution of eloquent function.

Direct electrical stimulation (DES) at the time of surgery allows assessment of eloquent function directly from the brain surface (invasive) and is considered the gold standard in brain mapping. Therefore, in order to determine the true clinical applicability of the non-invasive mapping technologies, this study proposes to: (1) assess the predictive value of fMRI and MEG for sensorimotor and language functions by comparing their results to DES and (2) determine whether fMRI or MEG provides the most consistent and accurate information. These aims will be accomplished by by co-registering all mapping data (invasive and non-invasive) in a modifiable 3D rendering. In this way, the DES to fMRI and MEG can be evaluated as well as fMRI to MEG compared. The rationale for the proposed research is that understanding the reliability of our current technology will allow for safer surgeries and preservation of neurologic function. The expected outcomes for the work proposed in Aims 1 and 2 are identification of a predictive value for fMRI and MEG and determination if one modality should be utilized over the other pre-operatively for the most accurate information. The results of this study are expected to have an important positive impact because identification of accurate pre-operative non-invasive mapping modalities will allow tailored testing and possibly lead to negation of the need for intra-operative mapping in certain cases. It will also enhance patient outcomes by improving patient safety. Furthermore, it will serve as the basis for a multi-institutional mapping data bank.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age equal to or greater than 19 years
* gender: male and female included
* brain tumor in or near an eloquent area of the brain that requires surgery
* benign or malignant intra-axial brain tumor
* primary or secondary intra-axial brain tumor
* appropriate body habitus for operating room positioning and airway protection for awake mapping
* appropriate mental status and capacity to participate with invasive or non-invasive mapping

Exclusion Criteria:

* any contraindication to MRI (i.e. implanted devices)
* inappropriate body habitus for safe positioning or airway protection
* no capacity to understand the study the study or consent to it
* significant disability precluding successful mapping
* positive pregnancy test in females
* end stage renal disease or severe renal dysfunction
* sleep apnea or any obstructive airway disease
* severe anxiety disorder
* metabolic encephalopathy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We propose enrolling 80 patients with brain tumors in or near eloquent brain regions who are appropriate candidates for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Location in the brain of the fMRI activations relative to intra-operative brain mapping | 5 years
  Assess the predictive value of fMRI for language and sensorimotor function by evaluating the location in the brain where the activity was found. The pre-operative locations will be compared to the intra-operative locations which are considered the gold standard. If the fMRI activations indicate the same gyrus/gyri as the intra-operative mapping, it is considered accurate. This is accomplished with special techniques integrating multiple data time points and types.
Location in the brain of the MEG activations relative to intra-operative brain mapping | 5 years
  Assess the predictive value of MEG for language and sensorimotor function by evaluating the location in the brain where the activity was found. The pre-operative locations will be compared to the intra-operative locations which are considered the gold standard. If the MEG activations indicate the same gyrus/gyri as the intra-operative mapping, it is considered accurate. This is accomplished with special techniques integrating multiple data time points and types.
Accuracy of fMRI and MEG in pre-operative brain mapping | 5 years
  Assess which mapping method provides the most consistent and accurate information in pre-operative mapping for language and sensorimotor function. Determination of the testing method that most often identifies the correct anatomic location of the eloquent function as dictated by the findings from outcomes 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Michele R Aizenberg Ansari, MD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No